CLINICAL TRIAL: NCT06574009
Title: Better Options for Chronic Cancer Pain: a SMART Study
Brief Title: Better Options for Chronic Cancer Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NURP-004-24S; I01CX002902-01 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain; Cancer Survivor; Opioid Dependence
Keywords: survivorship; chronic pain; analgesics
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Masking Description: Data analyst will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Multimodal pain care 9 months (Experimental): Findings from the comprehensive pain assessment will be used to inform an individualized, multimodal plan crafted by the team physician with the subject's collaboration
  Interventions: Behavioral: Multimodal pain care
- Medication optimization (Experimental): Findings from the comprehensive pain assessment will be used to inform a medication-focused pain plan.
  Interventions: Behavioral: Multimodal pain care; Device: Buprenorphine rotation
- Multimodal pain care 6 months / Opioid tapering 3 months (Experimental): Findings from the comprehensive pain assessment will be used to inform an individualized, multimodal plan crafted by the team physician with the subject's collaboration. After 6 mo, subjects will attempt to taper opioids
  Interventions: Behavioral: Multimodal pain care; Other: Opioid tapering
- Medication optimization 9 months (Experimental): Findings from the comprehensive pain assessment will be used to inform a medication-focused pain plan. Medications will be optimized following an algorithm the investigators created based upon NCCN's Survivorship Guidelines and AHRQ's comprehensive review of non-opioid treatments for chronic pain.
  Interventions: Drug: Medication optimization
- Medication optimization 6 months/ Buprenorphine rotation 3 months (Experimental): Findings from the comprehensive pain assessment will be used to inform a medication-focused pain plan. Medications will be optimized following an algorithm the investigators created based upon NCCN's Survivorship Guidelines and AHRQ's comprehensive review of non-opioid treatments for chronic pain. After 6mo, subjects will receive buprenorphine and attempt to taper opioids for following 3 mo.
  Interventions: Drug: Medication optimization; Device: Buprenorphine rotation
- Medication optimization 6 months/ Opioid tapering 3 months (Experimental): Findings from the comprehensive pain assessment will be used to inform a medication-focused pain plan. Medications will be optimized following an algorithm the investigators created based upon NCCN's Survivorship Guidelines and AHRQ's comprehensive review of non-opioid treatments for chronic pain. After 6mo, subjects will attempt to taper opioids for following 3 mo.
  Interventions: Drug: Medication optimization; Other: Opioid tapering

INTERVENTIONS:
Behavioral: Multimodal pain care — Behavioral therapy (as below), physical therapy, assistive devices (e.g. TENS, bracing), referrals to VA specialists (e.g. interventional pain), and complementary and integrative therapies (e.g. acupuncture or massage
  Arms: Medication optimization; Multimodal pain care 6 months / Opioid tapering 3 months; Multimodal pain care 9 months
Drug: Medication optimization — Medications will be optimized following an algorithm the investigators created based upon NCCN's Survivorship Guidelines and AHRQ's comprehensive review of non-opioid treatments for chronic pain.
  Arms: Medication optimization 6 months/ Buprenorphine rotation 3 months; Medication optimization 6 months/ Opioid tapering 3 months; Medication optimization 9 months
Device: Buprenorphine rotation — Subjects randomized to this arm at 6 months will be offered the chance to rotate from their full mu agonist opioid to buprenorphine using a standardized protocol
  Arms: Medication optimization; Medication optimization 6 months/ Buprenorphine rotation 3 months
Other: Opioid tapering — Subjects randomized to tapering will receive recommendations based upon the VA PBM's opioid tapering reference guide
  Arms: Medication optimization 6 months/ Opioid tapering 3 months; Multimodal pain care 6 months / Opioid tapering 3 months

SUMMARY:
This proposal is relevant to the 240,000 cancer survivors who continue to use opioids long after they have successfully completed treatment for cancer at the VHA, placing them at risk of opioid addiction and overdose, and other opioid-related problems. Yet, there are no programs at the VHA to help them find alternatives to opioids, nor evidence to inform the choice of interventions. This study will meet these needs by examining four interventions that are effective at reducing opioid use in patients with chronic musculoskeletal pain but have yet to be tested in cancer survivors on long term opioid therapy. The proposed work is relevant to the VHA Pain Office's mission to provide Veterans better pain management while limiting the risks of long-term opioid therapy and it aligns with VHA Research and Development's priority to examine clinical interventions for tapering opioids. Successful completion this project will keep VHA at the forefront of the battle against the opioid epidemic with a strategy that may be adapted to address the same needs in non-Veterans.

DETAILED DESCRIPTION:
Background: Twenty-four percent of Veterans who survive cancer remain on long term opioid therapy (LTOT) after completing cancer treatment, placing them at significant risk of opioid addiction, overdose, and other opioid-related health conditions. To reduce opioid use in this population, the investigators will examine the impacts of multimodal pain care and buprenorphine rotation - two strategies that have demonstrated efficacy in Veterans with musculoskeletal pain on LTOT but have not been tested in cancer survivors on LTOT, revealing a critical knowledge gap. The overall scientific premise of this project is that these two approaches can effectively reduce LTOT in cancer survivors without worsening chronic pain, and that they are better than pain medication optimization and opioid tapering. The primary objective is to examine which treatment strategy or combination of strategies is most successful at achieving a reduction in LTOT without worsening chronic pain over 6 and 9 months. The investigators will also identify the key challenges and strategies in the implementation of each treatment strategy to facilitate future translation of study findings into VA practice.

Significance: There are currently no care pathways at the VHA to help cancer survivors on LTOT find alternatives to opioids for managing chronic pain, nor evidence to guide which interventions to include. By addressing these unmet needs, this work aligns with POU-AMP's priority to examine clinical interventions for tapering opioid medications.

Innovation: The investigators are among the first to examine multimodal care and buprenorphine rotation to reduce LTOT in cancer survivors. Also, the investigators are among the first to apply VHA's evidence-based, stepped care model of multidisciplinary pain care to cancer survivors on LTOT.

Aim 1: To test if Veterans who receive multimodal pain care will be more likely to decrease total daily opioid use by at least 20% at 6 and 9 months without experiencing worsened pain interference compared to those who receive optimization of non-opioid pain medications.

Aim 2: To test if Veterans who do not respond to 6 months of multimodal care or medication optimization are more likely to achieve the desired outcome at 9 months when they are offered buprenorphine rotation as opposed to opioid tapering.

Exploratory Aim 3: To examine which combination of interventions is most likely to achieve the desired outcome at 9 months.

Aim 4: To understand the key challenges and strategies in the implementation of each intervention to facilitate future translation of study findings into practice.

Methodology: The investigators plan a two-site, two-stage, response-adaptive, comparative effectiveness trial following SMART (Sequential, Multiple-Assignment Randomized Trial) principles. The investigators will enroll 294 Veteran cancer survivors on LTOT who receive their care at the Indianapolis or Ann Arbor VAMC. Subjects will be randomized to either multimodal pain care or pain medication optimization at Stage 1. After 6 months, non-respondents will be randomized to buprenorphine rotation or opioid tapering in Stage 2. The primary outcome is a composite variable combining one objective outcome (opioid dose reduction) and one subjective outcome (pain interference), assessed at 6 and 9 months. The secondary outcomes are opioid dose reduction and pain interference individually.

Next Steps/Implementation: Successful execution of this project will provide actionable information, including an implementation strategy, that VHA's Offices of Pain Management and Oncology can put in place to support over 240,000 cancer survivors on LTOT for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Veterans must have had a qualifying solid tumor (bladder, breast, colorectal, head and neck, liver, lung, pancreas, prostate, or urinary tract) without evidence of active disease for at least 6 months
* Participants must be 6 months away from their last receipt of cytotoxic, radiation, or surgical cancer treatments but can be on hormonal or biologic therapies needed to sustain remission or cancer control.
* Participants must report pain >=4 (on 0-10 NRS) on their last 3 recordings in the electronic medical record. Veterans should be on Long Term Opioid Therapy (LTOT) defined as:

  * a qualifying opioid analgesic dispensed within the prior 30 days
  * plus 150 days' supply of a qualifying opioid (fentanyl, hydrocodone, hydromorphone, methadone, morphine, oxycodone, oxymorphone) in the 180 days before the most recent dispensing date with no between-fill gaps >40 days
* There must be advance agreement from their existing opioid prescriber to resume opioid prescribing after study

Exclusion Criteria:

* Veterans with total daily opioid doses >= 300 Morphine Milligram Equivalents (MME) will be excluded (higher doses require tapering prior to rotation to buprenorphine, which is something the investigators do not want to examine in this study)
* Veterans with referrals or visits to a substance abuse clinic within the prior 2 years will be excluded to avoid including individuals requiring addiction expertise that is not available one the multidisciplinary pain teams
* The investigators will also exclude Veterans with:

  * current or past use of buprenorphine
  * active alcohol use disorder or substance use
  * risk factors for opioid overdose (e.g. active suicidality or history of self-directed violence)
  * daily use of benzodiazepines
  * receipt of opioids from non-VA providers in the prior 3 months
  * or aberrant urine drug screen at baseline (cannabis is not exclusionary)
* To ensure the relevance of our work to as many Veteran cancer survivors as possible, the investigators will not exclude subjects meeting DSM criteria for opioid use disorder if their only source of opioids is the VA

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid dose reduction + Pain response (binary: yes/no) | 9 months
  The primary outcome is a composite variable which combines one objective outcome (opioid dose reduction) and one subjective outcome (pain interference) to reflect two outcomes of equal importance to Veterans. Veterans will be considered as achieving this outcome if they experience 20% reduction in opioid daily dose (in MEDD) from baseline and no worsening of pain interference by more than 1 point on the Pain Enjoyment of Life and General Activity (PEG) score.

SECONDARY OUTCOMES:
Opioid dose | 9 months
  total daily opioid dose will be measured in MEDD and based upon prescription tracking records and adjusted based upon self-report in the patient's diary.
Pain interference | 9 months
  Pain interference will be measured using PROMIS Pain Interference 6b measure
Pain intensity | 9 months
  Pain intensity will be measured using a 0-10 Numeric Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Maria J. Silveira, MD MA MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Karleen F Giannitrapani, PhD MA MPH, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No